CLINICAL TRIAL: NCT04475510
Title: Discontinuation of Antithrombotic Treatment Following Patent Foramen Ovale Closure in Young Patients With Cryptogenic Stroke. The HALTI Trial
Brief Title: Discontinuation of Antithrombotic Treatment Following Patent Foramen Ovale Closure in Young Patients With Cryptogenic Stroke
Acronym: HALTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Josep Rodes-Cabau (Other)
Responsible Party: Sponsor-Investigator, Josep Rodes-Cabau, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HALTI
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Patent Foramen Ovale; Ischemic Stroke; Bleeding Ulcer
Keywords: Transcatheter Patent Foramen Ovale (PFO) closure; Ischemic Stroke; Bleeding; Young patients
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke; Hemorrhage

STUDY DESIGN:
Intervention Model Description: At 12 months post-PFO closure, patients will discontinue the antiplatelet treatment. All patients will undergo a clinical evaluation and cerebral MRI at 12 months (before antiplatelet treatment cessation) and at 24 months post-PFO closure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antiplatelet treatment discontinuation (Experimental): At 12 months post-PFO closure, patients will discontinue the antiplatelet treatment. All patients will undergo a clinical evaluation and cerebral MRI at 12 months (before antiplatelet treatment cessation) and at 24 months post-PFO closure.
  Interventions: Other: Antiplatelet treatment discontinuation

INTERVENTIONS:
Other: Antiplatelet treatment discontinuation — All patients will undergo a clinical evaluation and cerebral MRI at 12 months (before antiplatelet treatment cessation) and at 24 months post-PFO closure.

SUMMARY:
To determine the safety of antithrombotic treatment discontinuation 12 months following successful transcatheter PFO closure.

DETAILED DESCRIPTION:
Young patients with a cryptogenic ischemic event undergoing transcatheter PFO closure exhibit a low but clinically relevant risk of bleeding (overall and major bleeding) at long-term follow-up, eventually exceeding the risk of ischemic events.

Importantly, the vast majority of major bleeding events seem to occur in patients receiving antiplatelet therapy. Preliminary data suggest that antiplatelet therapy discontinuation is not associated with any increase in ischemic events, and could potentially translate into a lower rate of major bleeding events at longer term follow-up. We therefore hypothesize that in young patients without any other comorbidities increasing the risk of stroke, shorter-term (≤1 year instead of lifelong) antiplatelet treatment could be a safe option following PFO closure.

ELIGIBILITY:
Inclusion Criteria:

* Successful transcatheter PFO closure with any approved device
* Patients ≤60 years diagnosed with a cryptogenic stroke/TIA who have undergone successful transcatheter PFO closure

Exclusion Criteria:

->60 year-old

* RoPE score <6
* Residual shunt ≥moderate following PFO closure
* Atrial fibrillation following PFO closure
* Presence of ≥2 cardiovascular risk factors (smoking, hypertension, dyslipidemia)
* Diabetes mellitus
* Thrombophilia (factor V Leiden, factor II mutation, anticardiolipin antibodies, lupus anticoagulant, anti-b2 glycoprotein-I antibodies, protein C deficiency, protein S deficiency)
* Recurrent cerebrovascular event (stroke, TIA) within the year following PFO closure
* Failure to provide signed informed consent
* Absolute contraindications for an MRI study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of new stroke events | 12 months
  1)Acute episode of a focal or global neurological deficit with at least one of the following: change in level of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopia, amaurosis fugax or other new neurological symptom(s) consistent with stroke.(2)Duration of a focal or global neurological deficit ≥ 24 hours OR < 24 hours if available neuroimaging documents a new hemorrhage or infarct; OR the neurological deficit results in death.
Presence of new ischemic lesions | 24-month follow-up
  Evaluated by MRI

SECONDARY OUTCOMES:
Number of new cerebral ischemic lesions | 24-month follow-up
  Evaluated by MRI
Volume of new cerebral ischemic lesions | 24-month follow-up
  Evaluated by MRI
Number of ischemic events | 24-month follow-up
  Stroke, TIA
Number of ischemic events | 3-year follow-up
  Stroke, TIA
Number of ischemic events | 4-year follow-up
  Stroke, TIA
Number of ischemic events | 5-year follow-up
  Stroke, TIA
Number of ischemic events | 6-year follow-up
  Stroke, TIA
Number of ischemic events | 7-year follow-up
  Stroke, TIA
Number of ischemic events | 8-year follow-up
  Stroke, TIA
Number of ischemic events | 9-year follow-up
  Stroke, TIA
Number of ischemic events | 10-year follow-up
  Stroke, TIA
Rate of bleeding | 24-month follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 3-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 4-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 5-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 6-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 7-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 8-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 9-year follow-up
  Life-threatening, major or minor bleeding
Rate of bleeding | 10-year follow-up
  Life-threatening, major or minor bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada